CLINICAL TRIAL: NCT05717764
Title: A Randomized, Open-label, Positive-controlled, Multicenter Phase Ш Study Comparing Mitoxantrone Hydrochloride Liposome Injection Combined With Capecitabine Versus Capecitabine Monotherapy in Patients With Recurrent Metastatic Nasopharyngeal Carcinoma Who Failed Platinum-containing Therapy
Brief Title: Clinical Study of Mitoxantrone Hydrochloride Liposome Injection Combined With Capecitabine Versus Capecitabine Monotherapy in Patients With Recurrent Metastatic Nasopharyngeal Carcinoma Who Failed Platinum-containing Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-031
Record Dates: First submitted 2023-01-11; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Recurrent Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will receive mitoxantrone hydrochloride liposome injection combined with capecitabine therapy
  Interventions: Drug: Mitoxantrone hydrochloride liposome injection; Drug: Capecitabine
- Control group (Active Comparator): Patients will receive capecitabine monotherapy.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome injection — Mitoxantrone hydrochloride liposome injection will be administered by intravenous infusion on day 1 in a 3-week treatment cycle.
  Arms: Experimental group
Drug: Capecitabine — Capecitabine will be administered orally in a 3-week treatment cycle, twice a day from day 1 to day 14 of each cycle.

SUMMARY:
This is a randomized, open-label, positive-controlled, multicenter Phase Ш study to evaluate the efficacy and safety of mitoxantrone hydrochloride liposome injection combined with capecitabine versus capecitabine monotherapy in patients with recurrent metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Five hundred patients with recurrent metastatic nasopharyngeal carcinoma will be randomly assigned to the experimental group or the control group. The experimental group will receive mitoxantrone hydrochloride liposome injection combined with capecitabine, and the control group will receive capecitabine alone. All patients will be treated until disease progression as determined by the investigator based on RECIST 1.1 criteria, intolerable toxicity, subject withdrawal of informed consent, initiation of new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first. Regular visits and imaging examinations will be conducted to compare the efficacy and safety of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and sign the informed consent form (ICF).
2. Age ≥ 18 years.
3. Nasopharyngeal carcinoma confirmed by histopathology.
4. Recurrent metastatic nasopharyngeal carcinoma that has previously failed treatment with first-line platinum-containing standard regimens and/or second-line standard regimens.
5. At least one evaluable lesion at baseline according to RECIST 1.1 criteria; The area should not have received previous radiotherapy, or there is evidence that the lesion has made definite progress after radiotherapy.
6. Eastern Cooperative Oncology Group (ECOG) score 0-1.
7. Toxic reaction caused by any previous antitumor treatment has recovered to grade 1 or below (except for alopecia, pigmentation, or other toxicities deemed by the investigator to pose no safety risk to the patient).
8. Adequate main organ function.
9. Female patients must have a negative blood HCG test (except for menopause and hysterectomy), Female patients of childbearing age and their partners must use effective contraception (For example: combination hormones [containing estrogen and progesterone] to suppress ovulation, progestogen contraception to suppress ovulation, intrauterine device, intrauterine hormone release system, bilateral tubal ligation, vasectomy, avoidance of sexual activity, etc) during the trial and within 6 months of the end of the last dose.
10. Male patients and their partners agree to use one of the contraceptive measures described in Article 9.

Exclusion Criteria:

1. Severe allergy to mitoxantrone or liposome; Previous severe, unexpected reactions to fluorouracil or known allergy to fluorouracil or to any excipients of capecitabine.
2. Previous treatment regimens containing capecitabine for recurrent or metastatic nasopharyngeal carcinoma; Patients with locally advanced nasopharyngeal carcinoma have previously experienced disease recurrence or metastasis during or within 6 months of use of capecitabine.
3. Patients with brain or meningeal metastasis.
4. Expected lifetime < 3 months.
5. Patients with active hepatitis B, hepatitis C or HIV.
6. Active bacterial infection, fungal infection, viral infection, or interstitial pneumonia requiring systemic therapy within 1 week prior to the first administration of the study drug.
7. Antitumor therapy such as chemotherapy, small-molecule inhibitors, immunotherapy (such as interleukin, interferon, or thymosin) within 4 weeks or 5 half-lives (whichever is shorter but at least 2 weeks) prior to initial administration of the study drug; Received Chinese patent drugs with antitumor activity within 14 days prior to administration.
8. Have received other investigational drugs within 4 weeks prior to initial administration.
9. Patients had major surgery within 3 months prior to initial dosing or plan to have major surgery during the study period.
10. Severe embolic events, such as cerebrovascular accidents (including transient ischemic attacks) and pulmonary embolism, occurred within 6 months prior to screening.
11. Other active malignant tumors within 2 years prior to the first study drug administration.
12. Abnormal heart function, including:

    Long QTc syndrome or QTc interval >480 ms; Complete left bundle branch block, second-degree or third-degree atrioventricular block; Severe, uncontrolled arrhythmias requiring medication; History of chronic congestive heart failure with NYHA ≥ grade 3; Cardiac ejection fraction less than 50% or lower than the lower limit of the laboratory test range within 6 months prior to screening; CTCAE version 5.0 ≥ grade 3 valvular heart disease; Uncontrolled hypertension (defined as measuring systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg when medically controlled); Myocardial infarction, unstable angina, history of severe pericardial disease, ECG evidence of acute ischemic or active conduction system abnormalities within 6 months prior to screening.
13. Prior treatment with doxorubicin or other anthracyclines and the cumulative doxorubicin doses greater than 350 mg/m^2 (anthracycline equivalent: 1 mg doxorubicin = 2 mg epirubicin = 2 mg daunorubicin = 0.5 mg normethoxydaunorubicin = 0.45 mg mitoxantrone).
14. Pregnant or lactating women.
15. Have any serious and/or uncontrollable medical conditions that, as determined by the investigator, may affect the patient's participation in the study.
16. Have severe gastrointestinal disorders that affect the ingestion, transport, or absorption of medications.
17. Other situations that the investigator determines to be inappropriate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the independent review committee (IRC) | Throughout the study period, up to approximately 2 years
  Progression-Free Survival PFS is defined as the time from randomization to progression or death
Overall survival (OS) | Throughout the study period, up to approximately 2 years
  Overall survival (OS) is defined as the duration from the date of diagnosis to death or last follow-up, with no restriction on the cause of death.

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed by the investigator and IRC | Throughout the study period, up to approximately 2 years
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to treatment
Disease control rate (DCR) assessed by the investigator and IRC | Throughout the study period, up to approximately 2 years
  Disease Control Rate (DCR) is defined as the percentage of patients who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents
Duration of Response (DOR) assessed by the investigator and IRC | Throughout the study period, up to approximately 2 years
  Duration of Response (DOR) is defined as time from the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death
Progression-free survival (PFS) assessed by the investigator | Throughout the study period, up to approximately 2 years
  Progression-Free Survival PFS is defined as the time from randomization to progression or death
Frequency and severity of AE (NCI CTCAE 5.0) | Throughout the study period, up to approximately 2 years
Blood concentrations of total and free mitoxantrone | At the end of Cycle 4 (each cycle is 28 days)

IPD SHARING:
Plan to Share IPD: No